

### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Breathing techniques and meditation during COVID-19 times for Health Care Workers

| 2020-0483 | |
|------------------------------|-----------------------|
| Study Chair: Santhosshi Nara | yanan |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

## STUDY SUMMARY

The goal of this research study is to learn if breathing techniques and meditation may help to reduce stress and improve lung health in health care workers during the COVID-19 pandemic.

### This study is investigational.

Meditation and breathing techniques may help manage your stress and may improve your lung health. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including time commitment.

You can read a list of potential risks below in the Possible Risks section of this consent.

Your participation in this study will last about 28 days.

The study will be performed at no cost to you.

You may choose not to take part in this study. You do not have to take part in this study, and your employment at MD Anderson will not be affected by your choice to

take part in this study or not.

#### 1. STUDY DETAILS

Signing this consent form does not mean that you will be able to take part in this study. You will first need to complete a screening questionnaire to help the study staff decide if you are eligible.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

If you are found to be eligible and you agree to take part in this study, you will be given access to a web-link with an instructional video about the breathing techniques and meditation. You are encouraged to perform the breathing techniques and meditation 2 times each day (1 time in the morning, and 1 time in the evening) for 28 days. Each session lasts about 5 minutes.

#### Each week:

- You will complete a questionnaire about your symptoms and quality of life. It should take less than 5 minutes to complete the questionnaire each time.
- You will measure how long you can hold your breath.

You will also complete a symptom questionnaire during Weeks 1 and 4. This should take about 10 minutes to complete each time.

#### 2. POSSIBLE RISKS

You should discuss the risks of **questionnaires** with the study chair. The known risks are listed in this form, but they will vary from person to person. Some questions may make you feel upset or uncomfortable. You may refuse to answer any question. If you have concerns after completing the questionnaire(s), you are encouraged to contact your doctor or the study chair.

It is recommended that you complete the questionnaires in a private setting and close your browser when you finish.

Your responses will be de-identified and linked to a study ID code, and will be kept in a secure data collection system. The study staff will consider your records confidential to the full extent permitted by law. Researchers will take appropriate steps to keep your information private. However, there is no guarantee of absolute privacy.

This study may involve unpredictable risks to the participants.

# 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

- 4. You may ask the study chair (Dr. Santhosshi Narayanan, at 346-228-6676 or SNarayanan2@mdanderson.org) or the study coordinator (Jewel Ochoa, at 713-563-4008 or jmochoa@mdanderson.org) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB - a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped at any time by the study chair or the IRB of MD Anderson.
- 7. MD Anderson may benefit from your participation and/or what is learned in this study.

# **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and/or shared with other researchers and/or institutions for use in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD

Anderson before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

# **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form
- B. Signing this consent and authorization form is optional but you cannot take part in this study if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer of MD Anderson at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to me. I have hit, ask questions, and talk about it with others as needed. I give permission to enroll me on this study. By signing this consent any of my legal rights. I will be given a signed copy of this cor | e the study chair<br>form, I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| The following signature line should only be filled out when the capacity to legally consent to take part in the study and/or her own behalf. | |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be per 2020-0483. | formed under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CFA witness signature is only required for vulnerable adult participants. If witness to assent page instruction of the witness to assent page instruction. | nessing the assent of a pediatric |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/orepresentative, using language that is understandable and apphave fully informed this participant of the nature of this study a risks and that the participant understood this explanation. | oropriate. I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

| <u>TRANSLATOR</u> | | |
|---|---|---|
| I have translated the above i | nformed consent as written (without a | dditions or |
| subtractions) into | and assiste | ed the people |
| • | lame of Language) | |
| obtaining and providing cons | ent by translating all questions and re | esponses during the |
| consent process for this part | icipant. | |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| 10 10 10 11 0 11 0 11 | | 57112 |
| Dlagge shock here if the t | ranalator was a mambar of the rassa | rob toom (If obsolved |
| | ranslator was a member of the resea<br>nslator, must sign the witness line belo | , |
| a williess, other than the trai | islator, must sign the withess line belt | Jvv.) |
| | TO THE VERBAL TRANSLATION | DATE |
| (OTHER THAN TRANSLATO | DR, PARENT/GUARDIAN, | |
| OR STUDY CHAIR) | | |

PRINTED NAME OF WITNESS TO THE VERBAL TRANSLATION